CLINICAL TRIAL: NCT04485975
Title: Preoperative Therapeutic Plasma Exchange and Surgical Treatment in Thyrotoxicosis Patients: a Single-centre Retrospective Cohort Study
Brief Title: Therapeutic Plasma Exchange in Thyrotoxicosis
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, İlker Murat Arer, Associate Professor Hakan Yabanoglu, Baskent University
Other Study IDs: KA20/244
Record Dates: First submitted 2020-06-30; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Thyrotoxicosis
MeSH Terms: conditions — Thyrotoxicosis | interventions — Plasma Exchange; Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Therapeutic plasma exchange — Therapeutic plasma exchange filtrates plasma and decreases thyroid hormone concentration in the blood
  Other Names: Thyroidectomy

SUMMARY:
Therapeutic plasma exchange (TPE) is indicated in cases where antithyroid medications cannot be used due to the side effects or attain no adequate hormonal suppression response at the highest dosage and in cases of rapid onset of clinical symptoms. This study presents the treatment results of patients who underwent TPE and subsequently operated for thyrotoxicosis.

DETAILED DESCRIPTION:
Background: Therapeutic plasma exchange (TPE) is indicated in cases where antithyroid medications cannot be used due to the side effects or attain no adequate hormonal suppression response at the highest dosage and in cases of rapid onset of clinical symptoms. This study presents the treatment results of patients who underwent TPE and subsequently operated for thyrotoxicosis.

Methods: The files of 27 patients who underwent preoperative TPE for thyrotoxicosis between January 1999 and February 2019 were retrospectively analyzed. The demographic and clinical features of the patients were included.

ELIGIBILITY:
Inclusion Criteria:

* thyrotoxicosis unresponsive to medication
* adverse reaction to the medications
* need for rapid treatment in patients that need urgent surgery

Exclusion Criteria:

* The patients who did not undergo surgery post-therapeutic plasma exchange
* Preoperative hypocalcemia,
* hemodynamically unstable patients
* patients not suitable for central catheter placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Therapeutic plasma exchange was performed in 27 thyrotoxic patients at the Adult Therapeutic Apheresis Center between January 1999 and February 2019. The patients were previously on treatment and follow-up in the Department of Endocrinology and Metabolism Diseases at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Thyroid hormone levels of patients after therapeutic plasma exchange | 1 week before the operation
  Concentration of serum thyroid hormone levels before thyroidectomy